CLINICAL TRIAL: NCT02771964
Title: Assessing Preoperative Falls as a Predictor for Postoperative Surgical Outcomes
Brief Title: Assessing Change in Patient-reported Quality of Life After Elective Surgery: an Observational Comparison Study
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Michael Avidan, Professor of Anesthesiology, Washington University School of Medicine
Other Study IDs: 201505035; UL1TR000448 (NIH); 1UH2AG050312-01 (NIH)
Record Dates: First submitted 2016-05-11; First posted 2016-05-13 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2019-01

CONDITIONS: Quality of Life; Surgical Procedure, Unspecified
Keywords: outcome assessment; postoperative period

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All patients: All patients receive both types of quality of life assessment, thus serving as their own controls.
  Interventions: Other: Quality of life survey

INTERVENTIONS:
Other: Quality of life survey — All enrolled patients complete a survey of baseline health during their visit to the preoperative assessment clinic and then complete a follow-up survey approximately 30 days after surgery.
  The intervention for this study is to compare self-reported quality of life ("How would you rate your quality of life now? (better/same/worse)") to the quantitative change in their VR-12 quality of life scores between the baseline survey and 30-day follow-up survey.

SUMMARY:
This study will compare two commonly-used methods for assessing patient-reported quality of life. The first is to assess quality of life before surgery and again after surgery using the same validated scale (ie Veterans Rand 12). The second is simply to ask patients whether or not they think their post-operative quality of life is better, worse, or the same. The investigators hypothesize that the second method may be inaccurate due to cognitive bias.

DETAILED DESCRIPTION:
All preoperative and postoperative quality of life data comes from the SATISFY-SOS (NCT02032030) surveys, which are administered to patients at the preoperative assessment visit and then approximately 30 days after surgery. To maximize the follow-up survey response rate, patients are emailed the survey (once), mailed hard copy surveys (two times), and phoned (up to five times).

The twelve items comprising the Veterans RAND 12 (VR-12) are items 24 through 35 on the survey, while the self-reported global quality of life question is item 1. The VR-12 is made up of two components: a physical component score (PCS), and a mental component score (MCS). Both scores are continuous on a scale from 0 to 100 (where higher is greater quality of life), and they are calibrated so that a score of 50 represents the US population mean (Kazis 2006, Selim 2009). The 30-day follow-up questionnaires also ask patients to self-report their change in quality of life. The question asks, "How would you rate your quality of life now?" with answer choices including "Better than before your procedure," "The same as before your procedure," and "Worse than before your procedure." Surgical specialty for the procedure is obtained from the electronic medical record. Using queries in MetaVision (iMDsoft, Needham, MA), the informaticist will provide the requested survey and medical record data to the investigators. He performs rigorous data validation on each queried variable.

SATISFY-SOS databases are hosted on a firewall-secured network server managed by the Department of Anesthesiology. The server is securely housed behind two locked doors within the departmental office suite and maintained and managed by the departmental IT team. Only the project Informaticist, Data Manager, and Director(s) have full access to these databases, which are also password-protected and encrypted for additional protection. Hardcopies of the baseline surveys are collected daily from the CPAP clinic and securely stored behind two locked doors within the Department of Anesthesiology. Baseline completed paper surveys are scanned into a digital image format (compressed TIFF). The digital image files are indexed and stored on a research file server that is attached to a private network with no public access. Survey email, mail and call lists are generated at Washington University in a similar manner to mailing lists for billing services. For each patient and date of service, a unique ID is generated and never duplicated. This unique ID is a nonsensical only meaningful to the research team.

Baseline surveys are processed by Solutions Data Systems. The digital image files are transmitted to Solutions Data Systems via secure file transfer protocol. When data entry has been confirmed, Solutions Data Systems deletes the digital image file from their servers. Press Ganey, a vendor specializing in patient survey distribution and collection, disseminates, collects, and processes 30-day and 1-year surveys. Paper surveys processed through automated scanning are all manually checked, and a manager listens to 10% of telephone surveys. All telephone surveys are recorded and available for future quality checks for performance improvement. Press Ganey stores the survey hardcopies for 90 days while the study team conducts spot-check quality assessments of the scanned data. The company then shreds the paper copies. Similarly, Press Ganey will hold copies of the electronic files and electronic recordings for 90 days, after which the electronic files are removed permanently from their system (and then only maintained by Washington University). During this 90-day period, the study team conducts additional quality assessments of the converted data.

Sample size considerations for this study were based on the primary outcome. The first component of the primary endpoint is comparing the median quality of life scores among the three self-reported change groups (better/same/worse). Using a minimum important difference of five points (Norman 2003), two tails, alpha of 0.05, and 80% power, the required sample size is 77 patients per group, or 231 total patients among the three groups. The second component of the primary outcome is the agreement between the two quality of life measures, as reflected by the kappa statistic. Kappa does not have sample size requirements beyond lack of sparse cells. The third component of the primary outcome is comparing the percentage agreement across the three different self-reported change groups. Since no studies have performed this type of comparison previously, the investigators pre-specified a 10% change as the minimum important change. Estimating 80% agreement, and using two tails, alpha=0.05, and 80% power, the required total sample size is 311 per group, or 933 total patients. Therefore, this study has adequate power for all of these endpoints.

The following statistical analyses will be performed, using alpha=0.05 and 95 percent confidence intervals, where appropriate. All analyses will be performed twice, once for VR-12 physical quality of life, and again for the VR-12 mental quality of life.

* Compare change in VR-12 QOL scores for those answering better/same/worse (Kruskal-Wallis). If significant, will use Wilcoxon Rank-Sum tests to compare each of the three groups, using a Bonferroni correction of alpha=0.017.
* Calculate overall agreement between the self-reported and validated quality of life measures (using weighted kappa, which penalizes disagreements in proportion to their seriousness).
* Calculate the overall percent of patients whose self-reported and validated quality of life scores matched (descriptive), including stratification by self-reported global change better/same/worse (compared using chi-square).
* Calculate the quality of life where an equal proportion of patients reported better and same quality of life (MCID for improvement), or same and worse quality of life (MCID for deterioration). This is an anchor-based approach (Wright 2012)
* Describe the change in VR-12 score and percent of patients reporting better, same, and worse quality of life for each of the following surgical specialties: neurosurgery, orthopedic, plastic, ophthalmologic, general, cardiac, gynecologic, otolaryngology, gastrointestinal/hepatobiliary, urologic, and "other."

Only those answering both the self-reported quality of life question and at least ten out of twelve VR-12 questions at baseline and 30 days will be included. The investigators will describe the characteristics of those with and without missing data. Multiple imputation will be used to fill in missing measurements for those missing two or fewer items on the VR-12 questionnaire.

ELIGIBILITY:
Inclusion Criteria: Age 18 or older, ability to read the English consent form, ability to consent, and plans to undergo elective surgery.

Exclusion Criteria: None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population is all adult patients undergoing elective surgery at Barnes Jewish Hospital who attend the center for preoperative assessment and planning.
Sampling Method: Non-Probability Sample
Enrollment: 17850 (Actual)
Dates: Start 2014-01; Primary Completion 2015-10 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Agreement between self-reported quality of life measurement (better/same/worse) and validated quality of life measurement (Veterans Rand 12 Item Health Survey) | Up to 4 months

SECONDARY OUTCOMES:
Minimum detectable difference in quality of life on the VR-12 scale, using self-reported quality of life (better/same/worse) as the anchor | Up to 4 months

OTHER OUTCOMES:
Change in quality of life across surgical specialties, using both the self-reported (better/same/worse) measure and the validated (VR-12) measure | Up to 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Avidan, MBBCh, Principal Investigator — Washington University School of Medicine
Locations (1):
- Department of Anesthesiology, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data can be provided upon email request.

REFERENCES:
- [Background] Kazis LE, Miller DR, Skinner KM, Lee A, Ren XS, Clark JA, Rogers WH, Sprio A III, Selim A, Linzer M, Payne SM, Mansell D, Fincke BG. Applications of methodologies of the Veterans Health Study in the VA healthcare system: conclusions and summary. J Ambul Care Manage. 2006 Apr-Jun;29(2):182-8. doi: 10.1097/00004479-200604000-00011. PMID 16552327
- [Background] Selim AJ, Rogers W, Fleishman JA, Qian SX, Fincke BG, Rothendler JA, Kazis LE. Updated U.S. population standard for the Veterans RAND 12-item Health Survey (VR-12). Qual Life Res. 2009 Feb;18(1):43-52. doi: 10.1007/s11136-008-9418-2. Epub 2008 Dec 3. PMID 19051059
- [Background] Norman GR, Sloan JA, Wyrwich KW. Interpretation of changes in health-related quality of life: the remarkable universality of half a standard deviation. Med Care. 2003 May;41(5):582-92. doi: 10.1097/01.MLR.0000062554.74615.4C. PMID 12719681
- [Background] Wright A, Hannon J, Hegedus EJ, Kavchak AE. Clinimetrics corner: a closer look at the minimal clinically important difference (MCID). J Man Manip Ther. 2012 Aug;20(3):160-6. doi: 10.1179/2042618612Y.0000000001. PMID 23904756
- [Derived] Kronzer VL, Jerry MR, Ben Abdallah A, Wildes TS, McKinnon SL, Sharma A, Avidan MS. Changes in quality of life after elective surgery: an observational study comparing two measures. Qual Life Res. 2017 Aug;26(8):2093-2102. doi: 10.1007/s11136-017-1560-2. Epub 2017 Mar 29. PMID 28357679
- See also: SATISFY-SOS registration — https://clinicaltrials.gov/ct2/show/NCT02032030